CLINICAL TRIAL: NCT01444391
Title: A Clinical Study of the Acclarent Tympanostomy Tube Delivery and Iontophoresis Systems In-Office
Brief Title: inVENT-visIOn Study
Acronym: inVENT-visIOn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005022
Record Dates: First submitted 2011-09-23; First posted 2011-09-30 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media
Keywords: Tympanostomy tube placement; iontophoresis
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tympanostomy Tube Placement (Experimental)
  Interventions: Device: Tympanostomy tube placement (Acclarent iontophoresis device)

INTERVENTIONS:
Device: Tympanostomy tube placement (Acclarent iontophoresis device) — Placement of tympanostomy tube by the Acclarent tympanostomy tube delivery system following delivery of anesthetic with Acclarent iontophoresis device

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the Acclarent Tympanostomy Tube Delivery System (TDS) for the placement of Tympanostomy Tube TT(s) under local anesthesia delivered by iontophoresis in an office/clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo tympanostomy tube insertion
* At least 6 months old
* Behavioral capacity and cooperative temperament to undergo an awake procedure (based on physician judgement)
* No history of sensitivity or reaction to anesthesia chosen for the procedure

Exclusion Criteria:

* Pregnant or lactating females
* Significantly atrophic, bimeric, or completely atelectatic tympanic membrane
* Otitis externa
* Lacerations or abrasions to the external auditory canal or damaged or denuded skin in the auditory canal
* Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane
* Electrically sensitive subjects and subjects with electrically sensitive support systems (pacemakers, defibrillators, etc.)
* Anatomy that precludes sufficient visualization of and access to the tympanic membrane
* Anatomy that necessitates tympanostomy tube placement in the posterior half of the tympanic membrane

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob W. Zeiders, M.D., Principal Investigator — South Coast Ear, Nose & Throat
Locations (1):
- South Coast Ear, Nose, & Throat, Port Saint Lucie, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tympanostomy Tube Placement
Started | 42
Completed | 41
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects including the lead-in subjects and the study cohort
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (26.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Procedural, Serious and Device-related Adverse Events.
Description: Adverse events which are procedural, serious, and device-related.
Time Frame: Procedure through 2 weeks post-procedure
Measure: Number; unit: subjects
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 42
subjects | 0

2. Primary Outcome: Device Success
Description: Device Success is defined as the successful delivery of the tympanostomy tube (TT) across the tympanic membrane (TM) using the Tube Delivery System(TDS). Device Success will be evaluated on a per device basis.
Time Frame: Day 0 (day of procedure)
Measure: Number; unit: devices
Units Other Than Participants: devices
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 42
Number analyzed (devices) | 63
devices | 55

3. Secondary Outcome: Procedure Success
Description: Procedure Success is defined as the successful placement of any tympanostomy tube in all enrolled ears in a given subject. Procedure Success is determined on a per subject basis.
Time Frame: Day 0 (day of procedure)
Measure: Number; unit: participants
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 42
participants | 42

4. Secondary Outcome: Procedure Tolerability
Description: Procedure Tolerability is defined as the proportion of subjects reporting the procedure as tolerable, where tolerable is defined as a score of 0 through 3, using the Wong-Baker FACES pain scale.The Wong-Baker FACES pain scoring system is a scale of 0 to 5, where 0 means 'no hurt', 1 = 'hurts a little bit', 2 = 'hurts little more', 3 = 'hurts even more', 4 = 'hurts whole lot' and 5 = 'hurts worst'. Procedure Tolerability will be determined on a per patient basis, with the patient's score being the average of the scores for the left and right ear if both ears are successfully treated with the Tube Delivery System.
Time Frame: Day 0 (day of procedure)
Population: The analysis population includes subjects with successful tube placement using the Tube Delivery System (TDS) in one or both ears. Six subjects were excluded for whom one ear had a successful TDS placement and one ear did not.
Measure: Number; unit: participants
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 36
participants | 36

5. Secondary Outcome: Tube Retention
Description: Tube retention is the presence of a tympanostomy tube placed successfully by the Tula TDS device across the tympanic membrane at the two-week follow-up visit.
Time Frame: 2 weeks post-procedure
Population: This outcome measure analysis includes evaluation only of ears with TDS-placed tube.
  Two subjects (3 ears) were excluded due to missing follow-up data. An additional 3 subjects (4 ears) were excluded because no TDS tube was placed. Three of the 37 participants analyzed had one of two study ears excluded, due to no TDS in that ear.
Measure: Number; unit: ears
Units Other Than Participants: ears
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 37
Number analyzed (ears) | 52
ears | 52

ADVERSE EVENTS:
Time Frame: Procedure (day 0) through 2 weeks post-procedure
Arm/Group | Tympanostomy Tube Placement
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 5/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanostomy Tube Placement (N=42)
Lymphoma - death (Blood and lymphatic system disorders) | 1 (1) — this event was not device or procedure-related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanostomy Tube Placement (N=42)
tube medialization (Ear and labyrinth disorders) | 2 (2)
occluded tube (Ear and labyrinth disorders) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1)
mild erythema at return electrode (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days